CLINICAL TRIAL: NCT00233337
Title: Open-label, Multi-center, Non-comparative Efficacy, Safety, and Tolerability Study of Co-artemether in the Treatment of Acute Uncomplicated Malaria in Non-immune Patients
Brief Title: Efficacy, Safety and Tolerability of Co-artemether in Non-immune Travelers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566A2401
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Acute Uncomplicated P. Falciparum Malaria
Keywords: Malaria, non-immune travelers
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: Co-artemether

SUMMARY:
This study will assess the safety and efficacy of co-artemether in the treatment of acute uncomplicated P. falciparum malaria in returning non-immune travellers

THIS STUDY IS NOT ENROLLING PATIENTS IN THE UNITED STATES

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for inclusion if they met all of the following criteria:

* Male or female aged 18 or older (prior to Amendment 1: more than 2 years old)
* Non-immune patients suffering from acute uncomplicated P. falciparum malaria, or mixed infection including P. falciparum, with parasitemia of less than or equal to 2% asexual P.falciparum parasites, confirmed by microscopy using Giemsa-stained thick film.
* Non-immune patients were regarded as those who had not spent the first five years of their life, nor the last five years in a malaria endemic area, and did not have acute P. falciparum malaria diagnosed during those past five years.
* Non-immune patients who had received prophylaxis with anti-malarials (excluding halofantrine) were included only if clear progression of acute P. falciparum infection was documented.
* Female patients were eligible to participate in the study if they were of non-childbearing potential or had a negative pregnancy test (urine or serum) at screening, and using an acceptable contraceptive method
* Patients, who had been informed of the study procedures and medication, and had given written informed consent and were willing to comply with the study protocol.

Exclusion Criteria:

* Patients were to be excluded from participation if they met any of the following criteria:

  * Known hypersensitivity to artemether or lumefantrine
  * Signs/symptoms indicative of severe/complicated malaria according to the WHO classification (e.g. cerebral malaria, see Post-text supplement 1)
  * Treatment with artemisinin derivatives within the previous 7 days
  * Concurrent administration of other treatment / prophylaxis for malaria
  * Concurrent administration of medications with potential hemolytic effects
  * Patients taking any drug metabolized by cytochrome isoenzymes CYP3A4 or CYP2D6
  * Received any other investigational drugs in the last 4 weeks before entry into the study
  * Severe cardiac impairment (i.e. evidence of existing cardiac conduction defect or overt symptoms of cardiac dysfunction or abnormalities of baseline ECG not associated with acute malaria); clinically relevant bradycardia or congestive cardiac failure with reduced left ventricular ejection fraction; pre-existing prolongation of the QT interval; history of symptomatic cardiac arrhythmias
  * Having received halofantrine or any other drug known to influence cardiac function within 4 weeks prior to Screening visit or taking other drugs that are known to prolong the QT interval, including class IA and III antiarrhythmics, neuroleptics, antidepressive agents, certain antibiotics (including some macrolides, fluoroquinolones, imidazole, and triazole antifungal agents), certain non-sedating antihistaminics (terfenadine, astemizole) and cisapride
  * History of splenectomy
  * Clinically significant abnormal baseline hematology (not associated with acute malaria) or clinical chemistry parameters, including evidence of hepatic or renal impairment, known disturbances of electrolyte balance e.g. hypokalemia or hypomagnesaemia
  * Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study, or concomitant disease which could mask the response to treatment
  * Unlikely, in the opinion of the investigator, to complete the dosing or follow-up periods, or who have evidence of alcohol, drug or solvent abuse.
  * Women who are pregnant, lactating or of childbearing potential and not using an acceptable contraceptive method were also excluded.

Other protocol inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients free of parasites in the blood after 28 days.

SECONDARY OUTCOMES:
Proportion of patients free of parasites in the blood after 7 days
Time to clearance of fever
Time to clearance of parasites in the blood
Proportion of patients with presence of sexual forms of the parasite in the blood (gametocytes);
Hematology and biochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals